CLINICAL TRIAL: NCT05227144
Title: An Open-label Phase 1b Study of ORIC-533 in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Study of ORIC-533 in Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ORIC Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ORIC-533-01
Record Dates: First submitted 2022-02-02; First posted 2022-02-07 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Relapsed or Refractory Multiple Myeloma
Keywords: CD73
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Interval 3+3 dose escalation design, followed by dose expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation (Experimental): ORIC-533 dosed orally, once per day of each consecutive 28-day cycle.
  Interventions: Drug: ORIC-533
- Dose Expansion (Experimental): RP2D dose
  Interventions: Drug: ORIC-533

INTERVENTIONS:
Drug: ORIC-533 — ORIC-533 once daily in consecutive 28-day cycles

SUMMARY:
The purpose of this study is to establish the Recommended Phase 2 Dose (RP2D), safety, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary antimyeloma activity of ORIC-533 in patients with multiple myeloma who have exhausted available treatment options

DETAILED DESCRIPTION:
ORIC-533 is a selective, orally bioavailable, small molecule inhibitor of CD73.This is an open-label, uncontrolled, multicenter, dose-finding study to assess the safety and preliminary antimyeloma activity of ORIC-533 in patients with relapsed or refractory multiple myeloma.

After the RP2D has been determined, dose expansion will further evaluate safety and preliminary antimyeloma activity of ORIC-533 in patients with relapsed or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma (MM) with relapsed or refractory disease according to IMWG Criteria
* Refractory to or not eligible for MM treatment regimens known to provide clinical benefit, including but not limited to an immunomodulatory agent, a proteasome inhibitor, and an anti-CD38 antibody, with documented disease progression
* Measurable disease at screening, including at least 1 of the criteria below:

  * Serum M-protein >0.5 g/dL (Patients with IgA myeloma in whom serum M protein is unreliable due to comigration of normal serum proteins may be considered eligible if total IgA >400 mg/dL)
  * Urine M-protein >200 mg/24 hours
  * Serum free light chains (FLC) assay: Involved FLC assay ≥10 mg/dL (≥100 mg/L) and an abnormal serum FLC ratio (<0.26 or >1.65)
  * Measurable bone or extramedullary plasmacytoma
* ECOG performance status ≤2
* Adequate bone marrow, renal, hepatic, pulmonary, and cardiac function defined as:

  * Estimated glomerular filtration rate ≥40 mL/min/1.73 m2.
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels both ≤3 times of upper limit of normal, unless there is suspected disease in the liver, in which case, no limit is set provided serum bilirubin is within eligibility criterion
  * Total bilirubin <1.5 × upper limit of normal (ULN), except in study participants with Gilbert's syndrome
  * Platelet count >40,000/μL
  * Absolute neutrophil count (ANC) >1000/μL
  * Left ventricular ejection fraction (LVEF) >45% as assessed by echocardiogram (ECHO) or multiple gated acquisition (MUGA)
  * Baseline oxygen saturation >92% on room air

Exclusion Criteria:

* Diagnosed or treated for another malignancy within 3 years prior to enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low risk prostate cancer after curative therapy
* Previous or concurrent plasma cell leukemia, AL amyloidosis, or POEMS (polyneuropathy, organomegaly, endocrinopathy, and skin changes) syndrome
* Known central nervous system (CNS) involvement
* Evidence of hyperviscosity syndrome
* Receiving any investigational treatment with a novel investigational agent (ie, no approved indication) within 28 days prior to the first dose of study drug
* Not recovered or stabilized from all toxicities from prior anticancer therapies and/or radiotherapy to Grade <2 with the exception of peripheral neuropathy
* Major surgery or radiation therapy within 14 days prior to first dose of study drug or incomplete recovery from adverse effects resulting from such procedure

  * Those who require limited course of radiation for management of bone pain for ≤14 days from initiation of therapy are not excluded
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days of starting therapy

  * Those who are on prophylactic antibiotics only, or on antibiotics and have confirmation of resolution of active infection, are eligible
* Daily requirement for corticosteroids (equivalent to >10 mg/day prednisone). Inhalation corticosteroids are exempt from this criterion

  * Exception: Corticosteroid dose equivalent >10 mg/day prednisone is acceptable if physiological levels require, so long as the dose is stable for at least 7 days prior to initiation of therapy
  * Lower amounts of corticosteroids that are not part of a daily requirement within 14 days prior to initiating therapy are also acceptable
* Known seropositive for active viral infection with human immunodeficiency virus (HIV), hepatitis B (HBV), or hepatitis C virus (HCV). Those who are seropositive because of hepatitis B vaccine are eligible. Patients who are positive for HBV core antibody or HBV surface antigen must have a negative polymerase chain reaction (PCR) result prior to enrollment. Those who are PCR positive will be excluded.
* History of class III or IV congestive heart failure or severe non-ischemic cardiomyopathy, unstable or poorly controlled angina, myocardial infarction, or ventricular arrhythmia within the previous 6 months of first dose of study drug
* QTcF >470 msec
* Other concurrent serious uncontrolled medical, psychological, or addictive conditions that, in the opinion of the investigator, may interfere with protocol compliance or contraindicates participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | 12 months
  RP2D as determined by interval 3+3 dose escalation design
Number of participants with adverse events | 36 months
  Safety and tolerability of ORIC-533
Number of participants with abnormal laboratory | 36 months
  Safety and tolerability of ORIC-533

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | 28 Days
  PK of ORIC-533
Area under the curve last concentration (AUClast) | 28 Days
  PK of ORIC-533
Elimination half-life (t1/2) | 28 Days
  PK of ORIC-533

CONTACTS AND LOCATIONS:
Overall Officials: Pratik S. Multani, MD, Study Director — ORIC Pharmaceuticals
Locations (8):
- United States (7):
  - James R. Berenson, MD, Inc., West Hollywood, California
  - Northside Hospital Cancer Institute, Atlanta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinical Rochester, Rochester, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The Charlotte-Mecklenburg Hospital Authority d/b/a Atrium Health, Charlotte, North Carolina
  - Swedish Health Services, Seattle, Washington
- Princess Margaret Cancer Research Center/University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No